CLINICAL TRIAL: NCT05486403
Title: The Appetite Toolbox: A Hybrid Type I Pilot Trial Testing the Effectiveness and Initial Implementation of a Programme Designed to Promote Children's Eating Regulation Skills in Preschool.
Brief Title: The Appetite Toolbox for Preschools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Keri McCrickerd, Research Scientist, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-169
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Eating Behavior; Self Regulation; Body Weight
Keywords: Hybrid Design; Preschool; Eating Behaviour; Appetite; Eating Regulation; Food intake
MeSH Terms: conditions — Feeding Behavior; Self-Control; Body Weight

STUDY DESIGN:
Intervention Model Description: The effectiveness measures are assessed using a parallel cluster-controlled design. The preschool center is considered a cluster for randomisation to either an Intervention Group or Waitlist Control Group. All preschool centers will deliver the Appetite Toolbox programme by the end of the research and contribute to the implementation outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Preschool Educators deliver the Appetite Toolbox programme directly to children over a period of six weeks after the pre-test and before the post-test effectiveness measures.
  Interventions: Behavioral: Appetite Toolbox Programme
- Waitlist Control (Other): Preschool Educators continue to deliver their usual preschool curriculum over a period of six weeks after the pre-test and before the post-test effectiveness measures. They will deliver the Appetite Toolbox programme directly to children after the post-test measures.
  Interventions: Behavioral: Appetite Toolbox Programme

INTERVENTIONS:
Behavioral: Appetite Toolbox Programme — Preschool educators are trained to deliver a bio-behavioural classroom-based programme focusing on building skills in i) appetite awareness, ii) attention/attention control and iii) sensing body cues. The programme is delivered using a combination of interactive story books, classroom props and activities, and mealtime transitions/routines.

SUMMARY:
This study uses a Hybrid research design to assess the effectiveness and implementation of a preschool-based programme - the Appetite Toolbox - delivered by Early Childhood Educators to promote children's appetite awareness and eating regulation skills. Children, their caregivers and classroom teachers will be recruited across 18 classrooms from preschool childcare centers. Preschool educators will deliver the Appetite Toolbox over a period of six weeks. Using a waitlist-control design we will measure changes in children's appetite awareness and eating regulation skills in school and describe implementation outcomes, such as fidelity, acceptability, and feasibility of the programme.

DETAILED DESCRIPTION:
The Appetite Toolbox is a programme developed for use in preschools and designed to promote children's appetite awareness and eating regulation skills through a series of books, classroom activities and mealtime routines developed with curriculum specialists and aligned to the Centre's core curriculum competencies (e.g. Language and Literacy, and Social and Emotional Development).

Using a Hybrid Type I cluster-controlled pilot design, the Appetite Toolbox for preschools study aims to:

i) Characterise the effectiveness of the Appetite Toolbox delivered over to increase children's awareness of appetite and eating regulation skills over a six-week period.

ii) Assess implementation of the Appetite Toolbox in preschool centers, with a focus on acceptability, appropriateness, fidelity, and feasibility of Appetite Toolbox as delivered by preschool educators.

The research team will also explore whether differences in home feeding practices and implementation factors moderated the effectiveness of the Appetite Toolbox in preschools.

Children will be recruited from N2, K1 and K2 classrooms across six preschools from the same anchor operator and three locations (18 classrooms in total, three per school). At each location, preschools will be randomised to complete the Appetite Toolbox programme over a period of six weeks, either immediately (intervention group) or later in the school year (waitlist-control group).

Effectiveness will be characterised by changes in children's ability to communicate meaningful changes in appetite, portion selections and tendency to snack in the absence of hunger. While implementation measures will assess the utility of training provisions alongside fidelity, acceptability, and appropriateness of the Appetite Toolbox programme in both the intervention and waitlist schools, captured through a series of questionnaires, in-class observations and interviews with teaching staff, central curriculum leaders and specialists.

The research results will provide important evidence for the impact and application of the Appetite Toolbox materials as a low-cost means to improve childhood eating behaviours via preschools and early years education, and inform the design of a larger-scale definitive trial.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Age 3 years 0 months to 6 years 11 months.
* English speaker (primary or secondary language)
* Enrolled in the childcare Program of the participating school

Parent/Legal guardian/Caregiver:

* Age 21 years and older
* English speaker (primary or secondary language)

Staff:

* Age 21 years and older
* English speaker (primary or secondary language)
* Currently employed as teaching staff at a participating preschool

Exclusion Criteria:

Children:

* Severe food allergy
* Does not normally eat the school's meal and snack provisions
* Non-English speaker (English is not primary or secondary language)
* A medical condition affecting appetite and metabolism

Parent/Legal guardian/Caregiver:

* Below 21 years old
* A non-English speaker (English is not primary or secondary language)

Staff:

* Below 21 years old
* A non-English speaker (English is not primary or secondary language)
* Not employed as teaching staff at a participating preschool

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 205 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Child appetite awareness | Baseline and Post-intervention (~6 weeks)
  Difference in accuracy in identifying changes in hunger and fullness pre- and post- meal for i) self (measured at lunch time), and ii) a fictional character described in a story. Ratings will be made on a custom 5-point picture rating scale ranging from "very hungry, my tummy is empty" (1) to "Very full, there is no room left in my tummy".
Child eating in the absence of hunger (EAH) | Baseline and Post-intervention (~6 weeks)
  Differences in the tendency for children to 'eat in the absence of hunger' (EAH) pre- and post-intervention. EAH is measured as the total calories consumed from a snack immediately presented within 10 minutes after consuming lunch, where more calories consumed confers greater EAH.

SECONDARY OUTCOMES:
Implementation outcomes (quantitative) | Baseline and Post-intervention (~6 weeks)
  Educator reported measures of appropriateness, acceptability and feasibility of the Appetite Toolbox programme, utility of the training and self-efficacy and intention to continue using the Appetite Toolbox resources. The implementation outcomes will be assessed using validated scales from Weiner and colleagues, with additional measures guided by the Consolidated Framework for Implementation Research (CFIR).
Implementation outcomes (qualitative) | Post-intervention (~6 weeks)
  A series of focus-group discussions will be held to capture further information on the implementation of the Appetite Toolbox programme. The focus group guides and subsequent coding will be guided by constructs outlined in the CFIR, including characteristics of the Appetite Toolbox programme (e.g. adaptability, perceived complexity), the preschool staff (e.g. knowledge, beliefs, self-efficacy) and organisational settings (e.g. learning climate, goals, priorities) .
Appetite Toolbox Fidelity | During the intervention (~ week 1, 2, 3, 4, 5, and 6 of the Appetite Toolbox programme)
  Educator fidelity to the Appetite Toolbox programme will be estimated using educator log-books and a classroom observation made by the research team, to characterise the use and delivery of the programme and meal transitions across classrooms.

OTHER OUTCOMES:
Child appetite traits | Baseline and Post-intervention (~6 weeks)
  Caregiver (home) reported child appetite traits, such as satiety responsivity, emotional overeating and slowness in eating, assessed using the Children's Eating Behaviour Questionnaire (CEBQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Institute for Clinical Sciences, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be made available upon reasonable request for research purposes, pending relevant approvals from the Institutional Review Board(s) and preschool organisation.